CLINICAL TRIAL: NCT04548713
Title: Control of Line Complications With KiteLock (CLiCK) in the Critical Care Unit
Brief Title: CLiCK in the Critical Care Unit
Acronym: CLiCK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Health (Other)
Collaborators: SterileCare Inc. (Industry); Center for Health Evaluation & Outcome Services (Unknown)
Responsible Party: Principal Investigator, Steve Reynolds, Critical Care Physician, Fraser Health
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0001
Record Dates: First submitted 2020-09-03; First posted 2020-09-14 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Central Venous Catheter Thrombosis; Central Venous Catheter Related Bloodstream Infection; Catheter Complications; Catheter Blockage; Catheter Dysfunction; Central Line-associated Bloodstream Infection (CLABSI); Catheter; Catheter Infection
Keywords: Ethylenediaminetetraaceticacid
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis

STUDY DESIGN:
Intervention Model Description: Multi-center, cluster-randomized, double-blinded, crossover study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4% EDTA CVC Lock (Experimental): Patients in this group will be given 4% EDTA as their CVC locking solution.
  Interventions: Device: 4% EDTA
- Standard of Care Saline CVC Lock (Active Comparator): Patients in this group will be given standard of care saline as their CVC locking solution.
  Interventions: Device: Saline

INTERVENTIONS:
Device: 4% EDTA — Sterile Catheter Lock Solution
  Other Names: KiteLock 4% Sterile Catheter Lock Solution
  Arms: 4% EDTA CVC Lock
Device: Saline — Saline Lock Solution
  Arms: Standard of Care Saline CVC Lock

SUMMARY:
Insertion of a central venous access device (CVAD) allows clinicians to easily access the circulation of a patient to administer life-saving interventions. Due to their invasive nature, CVADss are prone to complications such as infection, bacterial biofilm production, and catheter occlusion due to a thrombus. A CVAD is placed in up to 97% of patients in the intensive care unit, exposing this vulnerable population to risk of nosocomial infection and occlusion.

Current standard of care involves use of normal saline (for CVCs and PICCs) or citrate (for hemodialysis catheters) as a catheter locking solution. CVAD complications remain a problem with current standard of care.

4% tetrasodium Ethylenediaminetetraacetic acid (EDTA) fluid (KiteLock Sterile Locking Solution) possesses antimicrobial, anti-biofilm, and anti-thrombotic properties and is approved by Health Canada as a catheter locking solution. As such, it may be superior CVC locking solution than the present normal saline or citrate lock.

To our knowledge, the efficacy of an EDTA catheter locking solution has not yet been investigated in the intensive care patient population. Our team proposes to fill this knowledge gap by performing a multi-centre, cluster-randomized, crossover study evaluating the impact of KiteLock Sterile Locking Solution on a primary composite outcome of CLABSI, intraluminal occlusion, and alteplase use in the ICU of six ICU's compared to the standard of care saline lock.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age ICU/HAU Admission
* Presence of a central venous catheter requiring locking. This includes CVCs, IVADs, dialysis lines, and PICC lines.

Exclusion Criteria:

* Known or tested sensitivity to EDTA or edetate
* Confirmed or suspected pregnancy
* Patients who decline receiving blood products
* Physician, patient, or temporary substitute decision maker (TSDM) declines
* Currently enrolled in any other research study that may confound primary outcome measures. Co-enrollment in multiple studies will be considered on an individual basis
* Patients who were previously enrolled in the study. Patients who were enrolled in the first period are not eligible for (re-)enrolment in the second period, and patients who are enrolled in the study and transferred to another participating hospital are not eligible for (re-)enrollment at the receiving hospital. Patients who had been discharged from the unit to another hospital ward and are re-admitted to the critical care unit are no eligible for re-enrollment into the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1449 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Primary Composite Outcome of CVAD Complications Modifiable by Lock Procedures | From date of randomization until the date of catheter removal, ICU discharge, patient death death, or through study completion, an average of 9 months.
  incidence rate of the following: catheter obstruction requiring Alteplase, central-line associated bloodstream infection (CLABSI), or CVC replacement due to occlusion.

SECONDARY OUTCOMES:
Incidence rate of confirmed/suspected CLABSI | From date of randomization until the date of catheter removal, ICU discharge, patient death death, or through study completion, an average of 9 months
  Confirmed diagnosis of CLABSI as diagnosed by the patients healthcare team and on the patient chart.
Incidence rate of catheter occlusion requiring removal | From date of randomization until the date of catheter removal, ICU discharge, patient death death, or through study completion, an average of 9 months
  Confirmed occurrence of occlusion requiring removal as noted by the patients healthcare team and on the patient chart.
Incidence rate of catheter obstruction requiring alteplase use | From date of randomization until the date of catheter removal, ICU discharge, patient death death, or through study completion, an average of 9 months
  Confirmed obstruction requiring alteplase use as noted by the patients healthcare team and on the patient chart.
Direct cost related to alteplase use for catheter occlusion | through study From date of randomization until the date of catheter removal, ICU discharge, patient death death, or through study completion, an average of 9 months, an average of 16 months
  This outcome will be evaluated based on economical analysis.
Incidence rate of catheter-associated venous thrombosis | From date of randomization until the date of ICU discharge, patient death death, or through study completion, an average of 9 months
  Confirmed occurrence of catheter-associated venous thrombosis as noted by the patients healthcare team and on the patient chart.
Incidence rate of catheter colonization | From date of randomization until the date of catheter removal, ICU discharge, patient death death, or through study completion, an average of 9 months
  Confirmed occurrence of catheter colonization as noted by the patients healthcare team and on the patient chart.
Classification of microbial species isolated from colonized catheters | From date of randomization until the date of catheter removal, ICU discharge, patient death death, or through study completion, an average of 9 months
  A convenience sample of 15 colonized CVC's and 15 non-colonized CVC's (control) will be collected for further analysis as available.

OTHER OUTCOMES:
Subgroup analysis | From date of randomization until the date of catheter removal, ICU discharge, patient death death, or through study completion, an average of 9 months
  Those with their CVAD in place for 7 days or more will be analyzed in a separate subgroup for primary and secondary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Steven Reynolds, MD, Principal Investigator — Fraser Health
Locations (6):
- Canada (6):
  - Burnaby Hospital, Burnaby, British Columbia
  - Nanaimo Regional General Hospital, Nanaimo, British Columbia
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Surrey Memoral Hospital, Surrey, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ornowska M, Wong H, Ouyang Y, Mitra A, White A, Willems S, Wittmann J, Reynolds S. Control of Line Complications with KiteLock (CLiCK) in the critical care unit: study protocol for a multi-center, cluster-randomized, double-blinded, crossover trial investigating the effect of a novel locking fluid on central line complications in the critical care population. Trials. 2022 Aug 30;23(1):719. doi: 10.1186/s13063-022-06671-5. PMID 36042488